CLINICAL TRIAL: NCT03583879
Title: Using Gait Robotics to Improve Symptoms of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other); Assistive Technology Clinic, Canada (Other)
Responsible Party: Principal Investigator, Chris A. McGibbon, PhD, Professor, Faculty of Kinesiology, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPD001
Record Dates: First submitted 2018-06-28; First posted 2018-07-12 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; Dementia; Mild Cognitive Impairment
Keywords: Exoskeleton; Functional exercise
MeSH Terms: conditions — Parkinson Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exoskeleton exercise (Experimental): 8-week exercise program using the exoskeleton
  Interventions: Other: Exoskeleton exercise
- Standard exercise (Active Comparator): 8-week exercise program not using the exoskeleton
  Interventions: Other: Standard exercise
- No exercise (Placebo Comparator): 8-weeks of no treatment (wait-list control)
  Interventions: Other: No treatment

INTERVENTIONS:
Other: Exoskeleton exercise — Functional exercise with a robotic exoskeleton
  Arms: Exoskeleton exercise
Other: Standard exercise — Functional exercise without a robotic exoskeleton
  Arms: Standard exercise
Other: No treatment — Wait-list control
  Arms: No exercise

SUMMARY:
This study evaluates the benefits of exoskeleton-based exercise for improving mood and cognition in people with Parkinson's disease (PD). Participants with PD will be assigned one of three treatments delivered over 8-weeks: exoskeleton exercise (experimental intervention), non-exoskeleton exercise (active comparator), and wait-list control (no treatment).

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a movement disorder that significantly impairs mobility and increases risk of falls. Many people with PD also experience mild cognitive impairment (MCI) and some progress to Parkinson's disease dementia (PDD). Non-pharmacologic treatments such as physical activity and exercise are known to be neuroprotective and may improve cognition, mood and overall functioning in PD, but such interventions can be challenging for individuals with PD and cognitive impairment to fully participate in. Robotic over-ground exoskeletons have the potential to overcome this barrier; however there are no scientific data yet to support the use robotic exoskeletons in the PD population or those with mood disorder and/or declining cognitive function.

This therapeutic exploratory trial will fill this gap in knowledge and provide critical data for understanding how to integrate exoskeletons into clinical practice for age-related movement disorders when cognitive decline is present. Specifically we will test if an 8-week functional exercise program (gait, balance, aerobic exercise) using the KEEOGO Rehab(tm) exoskeleton can improve mood and cognition, as well as gait and balance, compared to the same functional exercise without using the exoskeleton, and a wait-list control (no treatment).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Cognitive function score >=16 on Montreal Cognitive Assessment (MoCA)
* Diagnosed with Parkinson's disease, Hoehn and Yahr stage 1 to 4
* Able to walk 10 meters without stopping and without human assistance (using assistive devices such as cane or walker if normally used)
* Waist and leg circumference and lower extremity lengths appropriate for a comfortable and safe fit in the KEEOGO device

Exclusion Criteria:

* Legally blind
* Treatment with another investigational drug or other intervention within the study period
* New medications started within last 4 weeks
* Skin condition that contraindicates use of orthotics or support braces
* Lower-extremity amputation above or below the knee
* Uncontrolled orthostatic hypotension
* Psychiatric disorders such as schizophrenia or bipolar disorder
* Other diagnosis that impairs gait and balance, such as, but not limited to, chronic obstructive pulmonary disease; peripheral arterial disease; vestibular disorders; cerebellar disease; cerebral palsy; muscular dystrophy; spinal cord injury; stroke or other brain injury; severe degenerative joint disease (osteoarthritis, rheumatoid arthritis, etc.)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | Baseline and 8 weeks
  10-item "Scales for Outcomes in Parkinson's-Cognition" (SCOPA-COG) instrument to evaluate cognitive function; Total score, range 0-43, higher scores = better cognitive functioning.
Change in mood | Baseline and 8 weeks
  14-item "Hospital Anxiety and Depression Scale" (HADS) instrument to measure mood disorder; Total score, range 0-42, higher scores = more severe mood disorder

SECONDARY OUTCOMES:
Change in UPDRS Mentation score | Baseline and 8 weeks
  "Unified Parkinson's Disease Rating Scale" (UPDRS), 4-item Section I - Mentation; Sub-scale score range 0-16, higher scores = worse symptoms.
Change in UPDRS Motor score | Baseline and 8 weeks
  "Unified Parkinson's Disease Rating Scale" (UPDRS), 14-item Section III - Motor; Sub-scale range 0-108, higher scores = worse symptoms.
Change in functional balance | Baseline and 8 weeks
  Brief version of Balance Evaluation Systems Test (Brief-BESTest) for balance, average of three tests.
Change in self-report balance confidence (of not falling) | Baseline and 8 weeks
  16 item "Activity-specific Balance Confidence" (ABC) for balance self-efficacy; Total score, 0-100, is average of items scaled on 0-100% confidence in doing specific tasks without falling, higher scores = better balance confidence
Change in gait speed | Baseline and 8 weeks
  Fast walking gait speed, average of three tests.
Change in dual-task gait cost index | Baseline and 8 weeks
  Dual-task gait cost index (DTGC); Calculated index score (0-1) based on ratio of gait speed during normal gait minus gait speed with cognitive distractor divided by normal gait speed, average of three tests.
Change in dual-task cognitive cost index | Baseline and 8 weeks
  Dual-task cognitive cost index (DTCC); Calculated index score (0-1) based on ratio of correct responses during sitting minus correct responses during gait divided by correct responses while seated, average of three tests.
Change in six minute walk test score | Baseline and 8 weeks
  Distance covered with 6 min walking, average of three tests

OTHER OUTCOMES:
Change in freezing of gait episodes | Baseline and 8 weeks
  6-item "Freezing of Gait Questionnaire" (FoG-Q) for measuring the impact of freezing of gait on mobility; Total score, range 0-24, higher scores = worse symptoms.
Change in physical function, pain, emotional well-being, and other indicators of health-related quality of life | Baseline and 8 weeks
  39-item "Parkinson's Disease health-related Quality of life" (PDQ-39) survey; Total score, 0-195, higher scores = worse health-related quality of life
Cumulative exercise dose | 2x per week for 8 weeks
  Actigraph activity monitor for quantifying cumulative energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Pearl Gryfe, Principal Investigator — Assistive Technology Clinic, Baycrest
Locations (2):
- Canada (2):
  - The University of New Brunswick, Fredericton, New Brunswick
  - Assistive Technology Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no individual participant data (IPD) sharing plan

REFERENCES:
- [Derived] McGibbon CA, Sexton A, Gryfe P. Exercising with a robotic exoskeleton can improve memory and gait in people with Parkinson's disease by facilitating progressive exercise intensity. Sci Rep. 2024 Feb 22;14(1):4417. doi: 10.1038/s41598-024-54200-y. PMID 38388571